CLINICAL TRIAL: NCT02486315
Title: Treatment of Coronary ARtery bIfurcation Narrowing by AXxess Stent Implantation
Acronym: CARINAX
Status: Completed | Type: Observational
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Carlo Briguori, MD, PhD, Clinica Mediterranea
Other Study IDs: NCTC005
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary bifurcation; coronary stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AXXESS stent: all consecutive patients with de novo bifurcation lesions treated at the Clinica Mediterranea (Naples) and at the "Sapienza" University (Rome) were screened for potential inclusion in the present study. Inclusion angiographic criteria were: 1) significant (≥70% diameter stenosis) bifurcation lesion; 2) MV reference diameter between 2.75 and 4.75 mm by visually estimated, 3) SB reference diameter ≥2.25 mm by visual estimate; 4) bifurcation angle (between the distal MV and the SB) <70° by visual estimate. Both protected and unprotected left main bifurcation lesions were allowed to be included, provided that all previous angiographic criteria were satisfied. Patients deemed eligible underwent AXXESS stent implantation
  Interventions: Device: AXXESS stent
- Control group: The control group is represented by patients with coronary bifurcation lesions treated with conventional techniques and standard balloon expandable drud eluting stents.
  This group was found retrospectively through a propensity score matching.

INTERVENTIONS:
Device: AXXESS stent — Axxess stent is a conically-shaped, self-expanding nitinol stent, with a 0.006-inch strut thickness, specifically designed to preserve and to match the anatomy of the bifurcation at the carina level. The stent is coated with Biolimus A9™, a highly lipophilic, semi-synthetic sirolimus analogue, immersed in the biodegradable polylactic acid (PLA) applied primarily to the abluminal surface. PLA completely dissolves after 6 to 9 months.The stent has 3 radiopaque markers at the distal end and one at the proximal end to aid in the visibility and placement. The AxxessTM stent is 7 Fr guiding catheter or Sheathless Guiding Catheter compatible. During the study period, the AxxessTM stent was available in 3 different diameters (3.0, 3.5 and 4.0 mm) and lengths (9, 10 and 14 mm)
  Groups: AXXESS stent

SUMMARY:
The Axxess™ Biolimus A9™ Eluting Coronary Bifurcation Stent System (AXXESS System; Biosensors, International, Morges, Switzerland) is a dedicated bifurcation stent, designed to cover the lesion at the level of the carina. Although deemed ideal for lesions involving only the proximal MV (1,0,0 according to Medina classification ref), this device may be used also in more complex bifurcation lesions when additional DES are required in the distal MV and/or in the SB. In the present registry the investigators report the performance and the efficacy of the self-expanding biolimus-eluting AxxessTM stent for the treatment of bifurcation lesions in a real-world population.

DETAILED DESCRIPTION:
Despite a comprehensive understanding of the physiological and technical issues regarding the coronary bifurcations lesions, percutaneous coronary intervention (PCI) in this setting remains challenging. When compared with non-bifurcation lesions, treatment of bifurcation lesions is associated with increased adverse clinical events and inferior angiographic outcomes including procedural complications. This is due to several technical challenges, including both anatomical (proximal-to-distal vessel mismatch [tapering], angulation and calcification) and procedural (plaque shift, and side-branch [SB] closure) features. Current balloon-expandable drug-eluting stent (DES) have not been designed to treat the bifurcation lesions; in particular, the inability of DES to adequately scaffold and preserve the ostium of SB represents a the major reason of failure, because this is the most common site for restenosis. Recently a large variety of dedicated bifurcation stents have been developed in order to 1) provide an easier access to the SB and to scaffold more effectively its ostium, and 2) adapt to main vassel (MV) tapering, and to the bifurcation anatomy.

ELIGIBILITY:
Inclusion Criteria:

1. significant (≥70% diameter stenosis) bifurcation lesion;
2. MV reference diameter between 2.75 and 4.75 mm by visually estimated
3. SB reference diameter ≥2.25 mm by visual estimate;
4. bifurcation angle (between the distal MV and the SB) <70° by visual estimate

Exclusion Criteria:

1. patients with contraindications to prolonged dual-antiplatelet therapy,
2. known sensitivity to "limus" compounds, stainless steel, titanium, or nickel;
3. inclusion in others studies on bifurcation lesions; and
4. all bifurcation lesions not satisfying the angiographic inclusion criteria reported above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients with de novo bifurcation lesions treated at the Clinica Mediterranea (Naples) and at the "Umberto I" University (Rome) were screened for potential inclusion in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
device success | intraprocedural
  successful deployment of the AxxessTM stent into the target lesion, without system failure or device-related complication.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Briguori, MD,PhD, Principal Investigator — Clinica Mediterranea

REFERENCES:
- [Background] Latib A, Colombo A. Bifurcation disease: what do we know, what should we do? JACC Cardiovasc Interv. 2008 Jun;1(3):218-26. doi: 10.1016/j.jcin.2007.12.008. PMID 19463303
- [Background] Wykrzykowska JJ, Grundeken MJ, Stankovic G, Di Mario C. Is there a need for dedicated devices? EuroIntervention. 2015;11 Suppl V:V139-42. doi: 10.4244/EIJV11SVA31. PMID 25983149
- [Background] Grube E, Buellesfeld L, Neumann FJ, Verheye S, Abizaid A, McClean D, Mueller R, Lansky A, Mehran R, Costa R, Gerckens U, Trauthen B, Fitzgerald PJ. Six-month clinical and angiographic results of a dedicated drug-eluting stent for the treatment of coronary bifurcation narrowings. Am J Cardiol. 2007 Jun 15;99(12):1691-7. doi: 10.1016/j.amjcard.2007.01.043. Epub 2007 May 7. PMID 17560877
- [Background] Buysschaert I, Dubois CL, Dens J, Ormiston J, Worthley S, McClean D, Ottervanger JP, Meredith I, Uren N, Wijns W, Whitbourn R, Mehran R, Lansky AJ, Bichalska M, Meis S, Verheye S. Three-year clinical results of the Axxess Biolimus A9 eluting bifurcation stent system: the DIVERGE study. EuroIntervention. 2013 Sep;9(5):573-81. doi: 10.4244/EIJV9I5A93. PMID 24058075
- [Background] Hasegawa T, Ako J, Koo BK, Miyazawa A, Sakurai R, Chang H, Dens J, Verheye S, Grube E, Honda Y, Fitzgerald PJ. Analysis of left main coronary artery bifurcation lesions treated with biolimus-eluting DEVAX AXXESS plus nitinol self-expanding stent: intravascular ultrasound results of the AXXENT trial. Catheter Cardiovasc Interv. 2009 Jan 1;73(1):34-41. doi: 10.1002/ccd.21765. PMID 19089934
- [Background] Garcia E, Unzue Vallejo L, Rodriguez-Rodrigo FJ. Placement of a single Axxess stent as new treatment strategy for Medina 1,0,0 left main stem bifurcation lesion. J Invasive Cardiol. 2014 Apr;26(4):E45-7. PMID 24717281
- [Background] Louvard Y, Thomas M, Dzavik V, Hildick-Smith D, Galassi AR, Pan M, Burzotta F, Zelizko M, Dudek D, Ludman P, Sheiban I, Lassen JF, Darremont O, Kastrati A, Ludwig J, Iakovou I, Brunel P, Lansky A, Meerkin D, Legrand V, Medina A, Lefevre T. Classification of coronary artery bifurcation lesions and treatments: time for a consensus! Catheter Cardiovasc Interv. 2008 Feb 1;71(2):175-83. doi: 10.1002/ccd.21314. PMID 17985377
- [Background] Lassen JF, Holm NR, Stankovic G, Lefevre T, Chieffo A, Hildick-Smith D, Pan M, Darremont O, Albiero R, Ferenc M, Louvard Y. Percutaneous coronary intervention for coronary bifurcation disease: consensus from the first 10 years of the European Bifurcation Club meetings. EuroIntervention. 2014 Sep;10(5):545-60. doi: 10.4244/EIJV10I5A97. PMID 25256198
- [Background] Medina A, Suarez de Lezo J, Pan M. [A new classification of coronary bifurcation lesions]. Rev Esp Cardiol. 2006 Feb;59(2):183. No abstract available. Spanish. PMID 16540043
- [Background] Noguchi T, Miyazaki MD S, Morii I, Daikoku S, Goto Y, Nonogi H. Percutaneous transluminal coronary angioplasty of chronic total occlusions. Determinants of primary success and long-term clinical outcome. Catheter Cardiovasc Interv. 2000 Mar;49(3):258-64. doi: 10.1002/(sici)1522-726x(200003)49:33.0.co;2-l. PMID 10700054
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Behan MW, Holm NR, Curzen NP, Erglis A, Stables RH, de Belder AJ, Niemela M, Cooter N, Chew DP, Steigen TK, Oldroyd KG, Jensen JS, Lassen JF, Thuesen L, Hildick-Smith D. Simple or complex stenting for bifurcation coronary lesions: a patient-level pooled-analysis of the Nordic Bifurcation Study and the British Bifurcation Coronary Study. Circ Cardiovasc Interv. 2011 Feb 1;4(1):57-64. doi: 10.1161/CIRCINTERVENTIONS.110.958512. Epub 2011 Jan 4. PMID 21205942